CLINICAL TRIAL: NCT01336972
Title: A Phase 2a, Single-center Study Investigating the Short-term Renal Hemodynamic Effects, Safety and Pharmacokinetics/ Pharmacodynamics of Oral Tolvaptan in Subjects With Autosomal Dominant Polycystic Kidney Disease at Various Stages of Renal Function
Brief Title: Short-term Renal Hemodynamic Effects of Tolvaptan in Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 156-09-284; 2010-019025-33 (EudraCT Number)
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A - eGFR > 60 ml/min/1.73m^2 (Experimental): Participants received tolvaptan for the first 3 weeks of the 6 week study. Participants were up-titrated on a weekly basis from tolvaptan 45/15 mg to 60/30 mg to 90/30 mg oral split-dose (AM and PM [8 hours later]) to the maximally tolerated dose.
  Interventions: Drug: Tolvaptan
- Group B - eGFR 30 to 60 ml/min/1.73m^2 (Experimental): Participants received tolvaptan for the first 3 weeks of the 6 week study. Participants were up-titrated on a weekly basis from tolvaptan 45/15 mg to 60/30 mg to 90/30 mg oral split-dose (AM and PM [8 hours later]) to the maximally tolerated dose.
  Interventions: Drug: Tolvaptan
- Group C - eGFR < 30 ml/min/1.73m^2 (Experimental): Participants received tolvaptan for the first 3 weeks of the 6 week study. Participants were up-titrated on a weekly basis from tolvaptan 45/15 mg to 60/30 mg to 90/30 mg oral split-dose (AM and PM [8 hours later]) to the maximally tolerated dose.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan was supplied as 15 and 30 mg tablets.
  Other Names: OPC-41061

SUMMARY:
The purpose of the trial was to determine the short-term effects of tolvaptan in patients with autosomal dominant polycystic kidney disease (ADPKD) at various levels of renal function.

DETAILED DESCRIPTION:
Renal function was assessed during screening with the estimated glomerular filtration rate (eGFR), which was calculated with the 4-variable modification of diet in renal disease (MDRD) equation using a minimum of 2 creatinine measurements. The eGFR values were used to categorize participants into 1 of 3 mutually exclusive strata (> 60 [Group A], 30 to 60 [Group B], and < 30 [Group C] mL/min/1.73 m^2). Each of the 3 groups received the same tolvaptan treatment.

During the 3-week treatment period, participants were up-titrated on a weekly basis from 45/15 mg to 60/30 mg to 90/30 mg (AM and PM [8 hours later] split-dose) to the maximally tolerated dose. The 3-week treatment period was followed by a 3-week post-treatment period during which no study medication was administered.

The effects of the highest tolerated split-dose of tolvaptan on renal hemodynamics and pharmacokinetic and pharmacodynamic parameters were assessed throughout the 6 weeks of the study. The reversibility of changes during the post-treatment period after withdrawal of the drug was determined and the acute transitory effects on kidney volume were also explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autosomal dominant polycystic kidney disease (ADPKD) by Ravine criteria.

Exclusion Criteria:

* Renal replacement therapy.
* Use of therapies for the purpose of affecting polycystic kidney disease (PKD) cysts.
* Evidence of significant renal disease, eg, active glomerular nephritides, renal cancer, single kidney.
* Significant risk-factors for renal impairment, eg, chronic use of diuretics, advanced diabetes, use of nephrotoxic drugs.
* History of significant coagulation defects or hemorrhagic diathesis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Czerwiec, MD, PhD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.; Ron T Gansevoort, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Boertien WE, Meijer E, de Jong PE, Bakker SJ, Czerwiec FS, Struck J, Oberdhan D, Shoaf SE, Krasa HB, Gansevoort RT. Short-term renal hemodynamic effects of tolvaptan in subjects with autosomal dominant polycystic kidney disease at various stages of chronic kidney disease. Kidney Int. 2013 Dec;84(6):1278-86. doi: 10.1038/ki.2013.285. Epub 2013 Jul 31. PMID 23903369
- [Background] Reddy B, Chapman AB. Acute Response to Tolvaptan in ADPKD: A Window to Predict Long-term Efficacy? Am J Kidney Dis. 2015 Jun;65(6):811-3. doi: 10.1053/j.ajkd.2015.03.004. No abstract available. PMID 26003607
- [Background] Boertien WE, Meijer E, de Jong PE, ter Horst GJ, Renken RJ, van der Jagt EJ, Kappert P, Ouyang J, Engels GE, van Oeveren W, Struck J, Czerwiec FS, Oberdhan D, Krasa HB, Gansevoort RT. Short-term Effects of Tolvaptan in Individuals With Autosomal Dominant Polycystic Kidney Disease at Various Levels of Kidney Function. Am J Kidney Dis. 2015 Jun;65(6):833-41. doi: 10.1053/j.ajkd.2014.11.010. Epub 2015 Jan 15. PMID 25600953
- [Background] Kramers BJ, van Gastel MDA, Boertien WE, Meijer E, Gansevoort RT. Determinants of Urine Volume in ADPKD Patients Using the Vasopressin V2 Receptor Antagonist Tolvaptan. Am J Kidney Dis. 2019 Mar;73(3):354-362. doi: 10.1053/j.ajkd.2018.09.016. Epub 2018 Dec 19. PMID 30578153
- [Derived] Chebib FT, Zhou X, Garbinsky D, Davenport E, Nunna S, Oberdhan D, Fernandes A. Tolvaptan and Kidney Function Decline in Older Individuals With Autosomal Dominant Polycystic Kidney Disease: A Pooled Analysis of Randomized Clinical Trials and Observational Studies. Kidney Med. 2023 Apr 14;5(6):100639. doi: 10.1016/j.xkme.2023.100639. eCollection 2023 Jun. PMID 37250503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 29 participants at one center in The Netherlands. Participants were stratified based on their estimated glomerular filtration rate (eGFR): >60, 30-60 and <30 millilitres (mL)/minute (min)/1.73 meter squared (m2). eGFR was assessed using the 4-variable modification of diet in renal disease (MDRD).
Pre-assignment Details: The trial consisted of a 2- to 42-day screening period, a 3-week treatment period, and a 3-week post treatment period.
Groups:
- eGFR > 60 mL/Min/1.73m2; eGFR 30-60 mL/Min/1.73m2; eGFR <30 ml/Min/1.73m2: Daily split-dose of tolvaptan titrated weekly to the maximally tolerated dose. Starting daily tolvaptan dose of 45mg/15mg titrated to 60mg/30mg, then 90mg/30mg based on tolerability.
Period: Overall Study
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 ml/Min/1.73m2
Started | 10 | 10 | 9
Completed | 9 | 9 | 9
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2 | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (7.1) | 47.8 (12.9) | 52.1 (6.7) | 46.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 2 | 14
  Male | 4 | 4 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Measured Glomerular Filtration Rate (mGFR) After 3 Weeks of Tolvaptan Treatment and at 3 Weeks Post Treatment.
Description: Renal function measurements were performed using the constant infusion method with 125I-iothalamate and 131I-hippuran. A priming solution containing 20 mL infusion solution (0.04 MBq of 125I-iothalamate and 0.03 MBq of 131I-hippuran) was given at 08:00 hours, followed by a constant infusion of 6 to 12 mL/h, with the lowest infusion rates in subjects with impaired renal function, based on previously known serum creatinine concentrations. Plasma concentrations of both tracers were allowed to stabilize during a 1.5-hour equilibration, which was followed by two 2-hour periods (09:30 to 11:30 hours and 11:30 to 13:30 hours) for simultaneous clearances of 125I-iothalamate and 131I-hippuran. Blood was drawn at 1, 2, 3, 4, and 5 hours post consumption of water/tolvaptan (08:30 hours). The mGFR was corrected for voiding errors.
Time Frame: After 3 weeks of treatment and 3 weeks post treatment
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 9 | 9 | 9
mL/min
  Final treatment change from Baseline | -8.0 (9.1) | -6.2 (6.2) | -0.7 (1.5)
  Post treatment change from Baseline | 0.1 (4.9) | -1.5 (4.0) | -1.2 (3.0)
Statistical Analysis 1: Comparison: eGFR > 60 mL/Min/1.73m2; A change of 10% was chosen as representing a clinically significant change in mGFR or ERPF. For this purpose, the alpha level was set at 0.05 and the beta level (power) at 95% instead of 80%, to decrease the chance of a false-negative finding; Test type: Superiority or Other; p < 0.05, paired t-test — Test to compare Final Treatment versus Baseline
Statistical Analysis 2: Comparison: eGFR 30-60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, paited t-test — Test to compare Final Treatment versus Baseline
Statistical Analysis 3: Comparison: eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Final Treatment versus Baseline
Statistical Analysis 4: Comparison: eGFR > 60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Post Treatment versus Baseline
Statistical Analysis 5: Comparison: eGFR 30-60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Post Treatment versus Baseline
Statistical Analysis 6: Comparison: eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Post Treatment versus Baseline
Statistical Analysis 7: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 8: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 9: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 10: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment
Statistical Analysis 11: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Mean Change From Baseline in Effective Renal Plasma Flow (ERPF) After 3 Weeks of Tolvaptan Treatment and at 3 Weeks Post Treatment.
Description: Renal function measurements were performed using the constant infusion method with 125I-iothalamate and 131I-hippuran. A priming solution containing 20 mL infusion solution (0.04 MBq of 125I-iothalamate and 0.03 MBq of 131I-hippuran) was given at 08:00 hours, followed by a constant infusion of 6 to 12 mL/h, with the lowest infusion rates in subjects with impaired renal function, based on previously known serum creatinine concentrations. Plasma concentrations of both tracers were allowed to stabilize during a 1.5-hour equilibration, which was followed by two 2-hour periods (09:30 to 11:30 hours and 11:30 to 13:30 hours) for simultaneous clearances of 125I-iothalamate and 131I-hippuran. Blood was drawn at 1, 2, 3, 4, and 5 hours post consumption of water/tolvaptan (08:30 hours).
Time Frame: After 3 weeks of treatment and 3 weeks post treatment
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 9 | 9 | 9
mL/min
  Final treatment change from Baseline | -16.9 (36.4) | -11.1 (18.4) | -1.7 (5.1)
  Post treatment change from Baseline | 4.3 (30.2) | -8.4 (17.7) | -1.3 (10.3)
Statistical Analysis 1: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Final Treatment versus Baseline for all treatment groups
Statistical Analysis 2: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Post Treatment versus Baseline for all treatment groups
Statistical Analysis 3: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 4: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 5: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment
Statistical Analysis 6: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment
Statistical Analysis 7: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment

3. Primary Outcome: Mean Change From Baseline in Filtration Fraction (GFR/ERFP) After 3 Weeks of Tolvaptan Treatment and at 3 Weeks Post Treatment.
Description: as for outcome 2
Time Frame: After 3 weeks of treatment and 3 weeks post treatment
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: Ratios
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 9 | 9 | 9
Ratios
  Final treatment change from Baseline | -0.005 (0.017) | -0.013 (0.016) | -0.010 (0.014)
  Post treatment change from Baseline | -0.003 (0.018) | 0.005 (0.015) | -0.016 (0.023)
Statistical Analysis 1: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Final Treatment versus Baseline
Statistical Analysis 2: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare Post Treatment versus Baseline for all treatment groups
Statistical Analysis 3: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 4: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 5: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 6: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment
Statistical Analysis 7: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment
Statistical Analysis 8: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment

4. Secondary Outcome: Mean Change From Baseline in Free Water Clearance After 3 Weeks of Tolvaptan Treatment and at 3 Weeks Post Treatment
Description: as for outcome 2
Time Frame: After 3 weeks of treatment and 3 weeks post treatment
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 9 | 9 | 9
mL/min
  Final treatment change from Baseline | 4.334 (3.268) | 2.822 (1.715) | 1.701 (1.225)
  Post treatment change from Baseline | -0.675 (1.475) | -0.195 (1.124) | 0.382 (0.543)
Statistical Analysis 1: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare Final Treatment versus Baseline for all treatment groups; Test type: Superiority or Other; p < 0.05, paired t-test
Statistical Analysis 2: Comparison: eGFR > 60 mL/Min/1.73m2; Test to compare Post Treatment versus Baseline; Test type: Superiority or Other; p > 0.05, paired t-test
Statistical Analysis 3: Comparison: eGFR 30-60 mL/Min/1.73m2; Test to compare Post Treatment versus Baseline; Test type: Superiority or Other; p > 0.05, paired t-test
Statistical Analysis 4: Comparison: eGFR <30 mL/Min/1.73m2; Test to compare Post Treatment versus Baseline; Test type: Superiority or Other; p < 0.05, paired t-test
Statistical Analysis 5: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney); Test to compare treatment groups at Final Treatment
Statistical Analysis 6: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test type: Superiority or Other; p > 0.05, paired t-test — Test to compare treatment groups at Final Treatment
Statistical Analysis 7: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Final Treatment
Statistical Analysis 8: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment
Statistical Analysis 9: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment
Statistical Analysis 10: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — Test to compare treatment groups at Post Treatment

5. Secondary Outcome: Time to Peak Plasma Concentration (Cmax) After 3 Weeks of Tolvaptan Treatment.
Description: Blood sampling for determination of tolvaptan concentrations took place at the Baseline, Final Treatment, and the Post Treatment or Early Termination visits.
  At the Final Treatment visit (Day 21 [+/- 1 day)]), blood samples were collected prior to the start of infusion of study treatment and at 1, 2, 3, 4, and 5 hours postdose.
  At the Baseline (Day 0), and Post Treatment visit (3 weeks [+/-3 days] after last dose), a blood sample was collected prior to the start of infusion of study treatment.
Time Frame: Day 0: 0 hour, Day 21: (0, 1, 2, 3, 4 and 5 hours postdose), 3 Weeks after last dose: 0 hour
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 8 | 9 | 9
ng/mL | 828 (297) | 591 (235) | 840 (355)

6. Secondary Outcome: Time to Peak Plasma Concentration (Tmax) After 3 Weeks of Tolvaptan Treatment.
Description: as for outcome 5
Time Frame: Day 0: 0 hour, Day 21: (0, 1, 2, 3, 4 and 5 hours postdose), 3 Weeks after last dose: 0 hour
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Median (Full Range); unit: hours
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 8 | 9 | 9
hours | 2.0 [1.00 to 3.00] | 2.0 [1.00 to 3.00] | 2.0 [1.00 to 5.00]

7. Secondary Outcome: Area Under the Concentration-time Curve From 0 to 5 Hours (AUC0-5) After 3 Weeks of Tolvaptan Treatment.
Description: as for outcome 5
Time Frame: Day 0: 0 hour, Day 21: (0, 1, 2, 3, 4 and 5 hours postdose), 3 Weeks after last dose: 0 hour
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 8 | 9 | 9
ng.h/mL | 2850 (774) | 2140 (863) | 3100 (1060)

8. Secondary Outcome: Percentage Change From Baseline in Total Kidney Volume (TKV) After 3 Weeks of Tolvaptan Treatment and at 3 Weeks Post Treatment.
Description: TKV was measured using magnetic resonance imaging.
Time Frame: After 3 weeks of treatment and 3 weeks post treatment
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 9 | 9 | 9
Percent
  Final treatment change from Baseline | -4.5 (3.7) | -4.6 (2.7) | -1.9 (1.9)
  Post treatment change from Baseline | -1.5 (2.3) | -2.4 (3.8) | -0.7 (2.5)
Statistical Analysis 1: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Comparison of all treatment groups versus Baseline at Final Treatment; Test type: Superiority or Other; p < 0.05, paired t-test
Statistical Analysis 2: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Comparison of all treatment groups versus Baseline at Post Treatment; Test type: Superiority or Other; p < 0.05, paired t-test
Statistical Analysis 3: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Mean Change From Baseline in 24 Hour Urine Volume After 3 Weeks Tolvaptan Treatment and at 3 Weeks Post Treatment.
Description: A 24-hour split urine sample (approximate times: 0700 to 1700 hours, 1700 hours to bedtime, and bedtime to 0700 hours) was collected beginning the day before the Baseline, Final Treatment, and Post Treatment visits and ending at admission to the renal function ward. Individual voids in a collection interval were pooled and the total volume determined.
Time Frame: 24 hours
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 9 | 9 | 9
mL
  Final treatment change from Baseline | 4551.1 (1792.7) | 3274.4 (1293.3) | 2215.0 (1142.0)
  Post treatment change from Baseline | -312.2 (468.2) | -287.2 (744.7) | 143.1 (390.4)
Statistical Analysis 1: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare Final Treatment versus Baseline for all treatment groups; Test type: Superiority or Other; p < 0.05, Paired t-test
Statistical Analysis 2: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare PostTreatment versus Baseline for all treatment groups; Test type: Superiority or Other; p > 0.05, Paired t-test
Statistical Analysis 6: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Mean Change From Baseline in 2 Hour Urine Volume After 3 Weeks Tolvaptan Treatment and at 3 Weeks Post Treatment.
Description: The volume of urine from each 2-hour urine collection in the renal function tests at Baseline, Final Treatment, and Post Treatment was recorded. Individual voids in a collection interval were pooled before determination of total volume.
Time Frame: 2 hours
Population: All participants who took any trial medication and had a postbaseline renal function test.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Number analyzed (Participants) | 9 | 9 | 9
mL
  Final treatment change from Baseline | 888.9 (730.3) | 625.6 (478.5) | 356.7 (283.2)
  Post treatment change from Baseline | -187.8 (218.2) | -10.0 (335.1) | 27.5 (155.0)
Statistical Analysis 1: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare Final Treatment versus Baseline for all treatment groups; Test type: Superiority or Other; p < 0.05, paired te-test
Statistical Analysis 2: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Final Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: eGFR > 60 mL/Min/1.73m2; Test to compare Post Treatment versus Baseline; Test type: Superiority or Other; p < 0.05, paired t-test
Statistical Analysis 6: Comparison: eGFR 30-60 mL/Min/1.73m2; Test to compare Post Treatment versus Baseline; Test type: Superiority or Other; p > 0.05, paired t-test
Statistical Analysis 7: Comparison: eGFR <30 mL/Min/1.73m2; Test to compare Post Treatment versus Baseline; Test type: Superiority or Other; p > 0.05, Paired t-test
Statistical Analysis 8: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR 30-60 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: eGFR 30-60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: eGFR > 60 mL/Min/1.73m2 vs eGFR <30 mL/Min/1.73m2; Test to compare treatment groups at Post Treatment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent to 7 days after the early termination visit or up to the 21 Day Post-Treatment Visit
Arm/Group | eGFR > 60 mL/Min/1.73m2 | eGFR 30-60 mL/Min/1.73m2 | eGFR <30 mL/Min/1.73m2
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 1/9
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | eGFR > 60 mL/Min/1.73m2 (N=10) | eGFR 30-60 mL/Min/1.73m2 (N=10) | eGFR <30 mL/Min/1.73m2 (N=9)
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | eGFR > 60 mL/Min/1.73m2 (N=10) | eGFR 30-60 mL/Min/1.73m2 (N=10) | eGFR <30 mL/Min/1.73m2 (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 5 | 5
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 3
Malaise (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 2 | 0 | 0
Thirst (General disorders) | 10 | 10 | 8
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin turgor decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 8 | 6 | 6
Polyuria (Renal and urinary disorders) | 9 | 9 | 7
Renal pain (Renal and urinary disorders) | 3 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Family stress (Social circumstances) | 0 | 1 | 0
Stress at work (Social circumstances) | 1 | 0 | 0
Fushing (Vascular disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No